CLINICAL TRIAL: NCT04909216
Title: Healthy Action Zone - Mindful Attention Training: A Mindfulness-Based Workshop for Firefighters
Brief Title: Mindful Attention Training Workshop for Firefighters
Acronym: HAZMAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Anka A Vujanovic, Associate Professor and Director of Graduate Education, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002213
Record Dates: First submitted 2021-05-19; First posted 2021-06-01 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Post Traumatic Stress Disorder; Mindfulness; Firefighters; Trauma; Mental Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Attention Workshop (Experimental): 50 participants will be randomized to the Mindful Attention Training (MAT) workshop. The 90-minute workshop will be conducted in group, online format.
  Interventions: Other: Mindful Attention Workshop
- Waitlist Control (No Intervention): 50 participants will be randomized to the waitlist control condition ("as usual" condition).

INTERVENTIONS:
Other: Mindful Attention Workshop — The 90-minute workshop will include a 15-minute break and include up to 15 participants. The workshop will be led by peer support staff, fire department psychologists, and/or fire department doctoral psychology practicum students. Each workshop will be facilitate by up to 3 workshop leaders. The workshop will provide (1) psychoeducation regarding common mental health concerns among firefighters, (2) introduction to the concept of mindful attention, why it is relevant to firefighters, and how it can prevent or decrease mental health symptoms, (3) 5 experiential mindful attention training exercises, and (4) discussion. Workshop co-leaders will teach 5 mindful attention exercises, and firefighters will practice each exercise and then engage in discussion about their experiences and provide feedback regarding the utility of the exercise for them personally and for firefighters, generally.
  Arms: Mindful Attention Workshop

SUMMARY:
The overarching goal of this study is to demonstrate the efficacy, feasibility, and acceptability of Mindful Attention Training (MAT), a novel mindfulness-based intervention that is specifically developed for firefighters. This project is designed to improve the health of firefighters, an integral, essential component of our national and international communities. Moreover, the study aims to promote health service psychologists by enhancing our contributions to the mental healthcare of firefighters, an understudied and underserved segment of the population by virtue of their service to our communities. This study therefore has significant potential to identify, develop, and promote an effective model of quality, evidence-based mental health promotion and illness prevention by integrating health service psychology into the fire service.

DETAILED DESCRIPTION:
Firefighters are repeatedly exposed to traumatic and stressful situations, increasing their vulnerability for the development of various psychological symptoms and disorders. As many as 32.4% of firefighters meet criteria for posttraumatic stress disorder (PTSD) with significantly more experiencing significant subclinical PTSD symptoms. Approximately 22% of firefighters are also at risk for depression, 46.8% reported serious suicidal ideation, and 15.5% reported having made a suicide attempt during heir firefighter tenure6. Alcohol use disorder (AUD) among firefighters is estimated at approximately 50%, nearly twice that of the general population.

Given the chronically stressful and potentially traumatic nature of the firefighting profession and the high rates of psychological disturbances among firefighters, the development of specialized mental health promotion and illness prevention programs for this vulnerable population is a priority. Mindfulness, generally defined as bringing one's full attention to the present moment and taking a stance of nonjudgmental acceptance to the ongoing flow of sensations, thoughts, and/or emotional states, has significant clinical relevance to the prevention and treatment of various psychological conditions. Mindfulness-based interventions have demonstrated efficacy with regard to various psychological symptoms, including PTSD, depression, and alcohol use. In a military context, mindful attention training has shown promise in terms of reducing the impact of combat on psychological health. However, no specialized mindfulness-based interventions exist for firefighters.

The overarching goal of this study is to demonstrate the efficacy, feasibility, and acceptability of Mindful Attention Training (MAT), a novel mindfulness-based intervention that is specifically developed for firefighters. This project is designed to improve the health of firefighters, an integral, essential component of our national and international communities. Moreover, the study aims to promote health service psychologists by enhancing our contributions to the mental healthcare of firefighters, an understudied and underserved segment of the population by virtue of their service to our communities. This study therefore has significant potential to identify, develop, and promote an effective model of quality, evidence-based mental health promotion and illness prevention by integrating health service psychology into the fire service.

Aim 1: To evaluate the efficacy of the Mindful Attention Training (MAT) workshop, as compared to waitlist comparison ("as usual" condition), on mental health promotion among firefighters, as defined by: self-reported levels of (1a) mindful attention and awareness, (1b) nonjudgmental acceptance, and (1c) nonreactivity at each time point.

Aim 2: To evaluate the efficacy of the MAT workshop, as compared to waitlist, on psychological 'illness' prevention among firefighters, as defined by: self-reported symptom severity of PTSD, depression, anxiety, suicidal ideation, and alcohol use at each time point.

Aim 3: To evaluate the feasibility and acceptability of the MAT workshop, as compared to waitlist, as defined by: (1) firefighters' self-reported helpfulness of the workshop and (2) firefighters' self-reported satisfaction ratings of the workshop.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Current employment as a firefighter with the Houston Fire Department

Exclusion Criteria:

* Persons who are not actively employed in the Houston Fire Department (e.g. former firefighters, retired firefighters)
* Current imminent risk of suicidality and/or homicidality (i.e., past month ideation with intent or plan)
* Inability to provide verbal or written consent
* Study personnel will not recruit or screen for individuals who fall into the following categories: pregnant women, prisoners, students for whom study personnel have direct access to/influence on grades, or economically and/or educationally disadvantaged persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Changes in mindfulness | Administered at each of the following timepoints: baseline, 1-week follow-up, 2-week follow-up, 1-month follow-up, 3-month follow-up, and 6-month follow-up
  To evaluate the efficacy of the Mindful Attention Training (MAT) workshop by examining self-reported levels of (1) nonjudgmental acceptance, (2) nonreactivity as well as (3) psychological resilience and (4) self-compassion at each time point using the following measure:
  - Five Facet Mindfulness Questionnaire (FFMQ; Baer et al., 2006): 39-item measure that assesses a participant's capacity for the following five factors: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience.
Changes in mindful attention | Administered at each of the following timepoints: baseline, 1-week follow-up, 2-week follow-up, 1-month follow-up, 3-month follow-up, and 6-month follow-up
  To evaluate the efficacy of the Mindful Attention Training (MAT) workshop by examining self-reported levels of mindful attention and awareness at each time point using the following measure:
  - Mindful Attention Awareness Scale (MAAS; Brown & Ryan, 2003): 15-item scale assessing a participant's capacity for mindful attention, a key component of mindfulness.
Changes in PTSD symptom severity | Administered at each of the following timepoints: baseline, 1-week follow-up, 2-week follow-up, 1-month follow-up, 3-month follow-up, and 6-month follow-up
  To evaluate the efficacy of the Mindful Attention Training (MAT) workshop on the symptom severity of PTSD at each time point using the following measure:
  - Posttraumatic Stress Disorder Checklist for the Diagnostic and Statistical Manual of Mental Disorders (PCL-5): 20-item self-report measure that assesses the 20 Diagnostic and Statistical Manual of Mental Disorders (DSM-5) symptoms of PTSD over the past month.
Changes in hazardous drinking patterns | Administered at each of the following timepoints: baseline, 1-week follow-up, 2-week follow-up, 1-month follow-up, 3-month follow-up, and 6-month follow-up
  To evaluate the efficacy of the Mindful Attention Training (MAT) workshop on the alcohol use and alcohol use severity at each time point using the following measure:
  - Alcohol Use Disorders Identification Test (AUDIT): 10-item screening measurement to assess any hazardous and harmful alcohol consumption during the past year.
Changes in depressive symptoms | Administered at each of the following timepoints: baseline, 1-week follow-up, 2-week follow-up, 1-month follow-up, 3-month follow-up, and 6-month follow-up
  To evaluate the efficacy of the Mindful Attention Training (MAT) workshop on the symptom severity of depression at each time point using the following measure:
  - Overall Depression Severity and Impairment Scale (ODSIS): 5 item measure assessing for past week depression-related symptoms.
Changes in suicidal thoughts | Administered at each of the following timepoints: baseline, 1-week follow-up, 2-week follow-up, 1-month follow-up, 3-month follow-up, and 6-month follow-up
  To evaluate the efficacy of the Mindful Attention Training (MAT) workshop on the severity and presence of suicidal thoughts at each time point using the following measure:
  - Beck Suicide Scale-5 (BSS-5): 5-item measure assessing the presence and intensity of suicidal thoughts.
Evaluate the feasibility and acceptability of the Mindful Attention Training (MAT) workshop | Administered at 1-week follow-up
  To evaluate the feasibility and acceptability of the MAT workshop, as compared to waitlist, as defined by: (1) firefighters' self-reported helpfulness of the workshop and (2) firefighters' self-reported efficacy ratings of the workshop using the following measure:
  - Post-MAT Workshop Questionnaire (Post-MAT): 10-item questionnaire assessing the degree to which participants found the workshop helpful and tolerable.
Changes in anxiety symptoms | Administered at each of the following timepoints: baseline, 1-week follow-up, 2-week follow-up, 1-month follow-up, 3-month follow-up, and 6-month follow-up
  To evaluate the efficacy of the Mindful Attention Training (MAT) workshop on the symptom severity of anxiety at each time point using the following measure:
  - Overall Anxiety Severity and Impairment Scale (OASIS): 5 item measure assessing for past week anxiety-related symptoms.

SECONDARY OUTCOMES:
Evaluate group dynamics | Administered at 1-week follow-up
  To evaluate the group dynamics of the MAT workshop using the following measure:
  - Group Evaluation Scale (GES; Joyce, 2005): 7-item measure assessing how the participant felt while participating in the group, particularly comfortability and sense of being understood by other group members.
Evaluate group cohesion | Administered at 1-week follow-up
  To evaluate the cohesion of each group in the MAT workshop using the following measure:
  - Group Cohesion Questionnaire (GCQ; MacKenzie, 1983): 12-item measure assessing a participant's view of the cohesion of the group and the quality of the group dynamic.
Evaluate occupational stress | Administered at each of the following timepoints: baseline, 1-week follow-up, 2-week follow-up, 1-month follow-up, 3-month follow-up, and 6-month follow-up
  To evaluate the influence of the Mindful Attention Training (MAT) workshop on self-reported occupational stress levels at each time point using the following measure:
  - The Sources of Occupational Stress (SOOS-14): 14-item self-report measure used to assess levels of occupational stress (i.e., harmful physical and psychological responses that occur when job requirements do not align with the worker's abilities, resources, and/or needs) among firefighters.

CONTACTS AND LOCATIONS:
Locations (1):
- Trauma and Stress Studies Center, Houston, Texas, United States